CLINICAL TRIAL: NCT06096181
Title: A Prospective Study Comparing Total Intravenous Anesthesia With Propofol and Remifentanil vs. Propofol and Dexmedetomidine in Adolescent Idiopathic Scoliosis Patients Undergoing Posterior Spinal Fusion and Instrumentation
Brief Title: Propofol + Remifentanil vs. Propofol + Dexmedetomidine in Adolescent Idiopathic Scoliosis Patients Having Spine Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary surgeon decided to prematurely halt the study because he anecdotally felt that one of the trial drugs (Dexmedetomidine) could affect the motor evoked potential monitoring necessary for the surgery.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Glenn Tan, M.D., Director of Pediatric Anesthesia, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00002614
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-08

CONDITIONS: Adolescent Idiopathic Scoliosis; Multimodal Analgesia; Opioid Induced Hyperalgesia; Remifentanil; Dexmedetomidine; Posterior Spinal Fusion
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The following persons are masked:
  1. Participant and parents
  2. Pediatric Intensive Care Unit (PICU) staff taking care of patient postoperatively
  3. Surgeon
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propofol + Remifentanil (Active Comparator): Participants are randomly selected to receive Propofol + Remifentanil TIVA as their anesthesia. Dose of IV Propofol is 100-200 mcg/kg/min and dose of Remifentanil is 0.2-0.5 mcg/kg/min. TIVA is titrated to keep bispectral index (BIS) < 55-60 to ensure patient is asleep.
  Interventions: Drug: Remifentanil TIVA; Drug: Propofol TIVA
- Propofol + Dexmedetomidine (Active Comparator): Participants are randomly selected to receive Propofol + Dexmedetomidine as their anesthesia. Dose of Propofol is 100-200 mcg/kg/min and dose Dexmedetomidine is ) 0.2-0.7 mcg/kg/hr. TIVA is titrated to beep bispectral index (BIS) < 55-60 to ensure patient is asleep.
  Interventions: Drug: Dexmedetomidine TIVA; Drug: Propofol TIVA

INTERVENTIONS:
Drug: Remifentanil TIVA — Remifentanil is more commonly used in the TIVA combination for pediatric patients having this surgery.
  Other Names: Ultiva TIVA
  Arms: Propofol + Remifentanil
Drug: Dexmedetomidine TIVA — Dexmedetomidine is less commonly used in the TIVA combination for pediatric patients having this surgery.
  Other Names: Precedex TIVA
  Arms: Propofol + Dexmedetomidine
Drug: Propofol TIVA — Propofol is an anesthetic drug that causes sleep during surgery.
  Other Names: Diprivan TIVA

SUMMARY:
Patients with Adolescent Idiopathic Scoliosis may need surgery to correct their scoliosis. General anesthesia is required for this surgery, and a multimodal analgesic regimen using combinations of opioid and non-opioid medications is the standard of care. The purpose of this study is to compare two combinations of total intravenous anesthetic medications in children with Adolescent Idiopathic Scoliosis having posterior spinal fusion surgery.

Participants in the study will be randomly selected to receive either Propofol and Remifentanil or Propofol and Dexmedetomidine as their total intravenous anesthesia (TIVA). TIVA is favored over gas anesthesia because gas anesthesia can affect the neurological monitoring necessary for this surgery.

The first combination (Propofol + Remifentanil) is the most common one used for this surgery at our institution, and the second combination (Propofol + Dexmedetomidine) is more commonly used in adult spine surgery. Though Dexmedetomidine is not approved for pediatric use by the FDA, it is widely used in pediatric patients for procedural sedation and surgical anesthesia in the US and worldwide. Both anesthetic combinations are used safely in adult and pediatric patients at our institution.

Although remifentanil works fast and is an excellent pain medication during surgery, there are reports that it's use can cause increased pain sensitivity and greater need for narcotic pain medication after surgery. This phenomenon is known as opioid-induced hyperalgesia. The investigators hypothesize that avoiding the use of remifentanil in the TIVA by using dexmedetomidine could avoid OIH and thus result in superior postop pain control.

Our study's primary goal is to measure the total opioid consumption on postoperative days (POD)# 0 and 1. Our secondary goals are to measure the pain scores on a visual analog scale (VAS) on POD# 0 and 1, measure the time it takes for participants to move their feet to command when surgery is done, and measure the time it takes for participants to be extubated when surgery is done. By comparing these measurements, the investigators hope to find out if there is any significant difference between the two TIVAs in terms of postop opioid requirements, pain scores, and time to wake up from anesthesia.

The investigators hope that our study gives us more knowledge on how to better treat postoperative pain in children who have spine surgery to correct their

DETAILED DESCRIPTION:
Patients with Adolescent Idiopathic Scoliosis (AIS) may need surgery to correct their scoliosis. General anesthesia is required for this surgery, and a multimodal analgesic regimen using combinations of opioid and non-opioid medications is the standard of care. Total intravenous anesthesia (TIVA) is the usual anesthetic technique of choice.

The purpose of this study is to compare two combinations of TIVA medications in children AIS having posterior spinal fusion surgery.

The most common TIVA for this surgery at our institution is Propofol + Remifentanil. Remifentanil is a popular choice because of its rapid onset, extremely short context-sensitive half-life, potency, and its rapid recovery from drug effect. However, an important concern with intraoperative remifentanil infusion is the possible development of acute opioid-induced hyperalgesia (OIH). In adults, OIH is a well-documented feature linked to intraoperative remifentanil administration, manifesting as increased postoperative analgesic requirement and paradoxical increase in sensitivity to painful stimuli. In pediatric patients, the phenomenon is not as well characterized.

An alternative TIVA that is very commonly used for adult spine surgery is propofol + dexmedetomidine (DEX). DEX is a highly selective alpha2-adrenergic receptor agonist with sedative, analgesic, and sympatholytic properties.

Despite the lack of FDA approval for pediatric use, DEX is widely used off-label in pediatric patients in the US and worldwide and has previously been shown to be safe and efficacious for various clinical indications including procedural sedation, craniotomy-awake-surgery, cardiac surgery, and posterior spinal fusion for scoliosis. DEX is currently used safely in pediatric and adult spine patients in our institution. The most common adverse effect is intraoperative bradycardia.

Participants will be randomized to receive one of the two TIVAs to see if one or the other results in lower opioid consumption, and lower Visual Analog Scale (VAS) pain scores in the post-operative period (POD# 0 and 1). The investigators hypothesize that the use of DEX will avoid OIH and this will lead to less opioid consumption in the postoperative period, and superior postoperative pain control. The investigators also hope to show that the use of DEX will not significantly prolong time to moving feet to command and extubation at conclusion of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years old
* American Society of Anesthesiology Physical Status Classification (ASA Class) 1 and 2
* Have diagnosis of Adolescent Idiopathic Scoliosis
* Undergoing Posterior Spinal Fusion with instrumentation for scoliosis correction
* Matched on age, sex, and the number of vertebral levels fused

Exclusion Criteria:

* Neuromuscular scoliosis
* Allergy to any of the multi-modal analgesia regimen drugs
* Use of serotonergic drugs, monoamine oxidase inhibitors (MAOI), mixed agonist/antagonist opioid analgesics

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Tan, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young CD, McLuckie D, Spencer AO. Anaesthetic care for surgical management of adolescent idiopathic scoliosis. BJA Educ. 2019 Jul;19(7):232-237. doi: 10.1016/j.bjae.2019.03.005. Epub 2019 May 14. No abstract available. PMID 33456896
- [Background] Lee CS, Merchant S, Chidambaran V. Postoperative Pain Management in Pediatric Spinal Fusion Surgery for Idiopathic Scoliosis. Paediatr Drugs. 2020 Dec;22(6):575-601. doi: 10.1007/s40272-020-00423-1. Epub 2020 Oct 23. PMID 33094437
- [Background] Gall O, Aubineau JV, Berniere J, Desjeux L, Murat I. Analgesic effect of low-dose intrathecal morphine after spinal fusion in children. Anesthesiology. 2001 Mar;94(3):447-52. doi: 10.1097/00000542-200103000-00014. PMID 11374604
- [Background] Goodarzi M. The advantages of intrathecal opioids for spinal fusion in children. Paediatr Anaesth. 1998;8(2):131-4. doi: 10.1046/j.1460-9592.1998.00737.x. PMID 9549739
- [Background] Eschertzhuber S, Hohlrieder M, Keller C, Oswald E, Kuehbacher G, Innerhofer P. Comparison of high- and low-dose intrathecal morphine for spinal fusion in children. Br J Anaesth. 2008 Apr;100(4):538-43. doi: 10.1093/bja/aen025. Epub 2008 Feb 27. PMID 18305080
- [Background] Tripi PA, Poe-Kochert C, Potzman J, Son-Hing JP, Thompson GH. Intrathecal morphine for postoperative analgesia in patients with idiopathic scoliosis undergoing posterior spinal fusion. Spine (Phila Pa 1976). 2008 Sep 15;33(20):2248-51. doi: 10.1097/BRS.0b013e31817bd8be. PMID 18794769
- [Background] Ibach BW, Loeber C, Shukry M, Hagemann TM, Harrison D, Johnson PN. Duration of intrathecal morphine effect in children with idiopathic scoliosis undergoing posterior spinal fusion. J Opioid Manag. 2015 Jul-Aug;11(4):295-303. doi: 10.5055/jom.2015.0278. PMID 26312956
- [Background] Ross AK, Davis PJ, Dear Gd GL, Ginsberg B, McGowan FX, Stiller RD, Henson LG, Huffman C, Muir KT. Pharmacokinetics of remifentanil in anesthetized pediatric patients undergoing elective surgery or diagnostic procedures. Anesth Analg. 2001 Dec;93(6):1393-401, table of contents. doi: 10.1097/00000539-200112000-00008. PMID 11726413
- [Background] Donmez A, Kizilkan A, Berksun H, Varan B, Tokel K. One center's experience with remifentanil infusions for pediatric cardiac catheterization. J Cardiothorac Vasc Anesth. 2001 Dec;15(6):736-9. doi: 10.1053/jcan.2001.28319. PMID 11748523
- [Background] German JW, Aneja R, Heard C, Dias M. Continuous remifentanil for pediatric neurosurgery patients. Pediatr Neurosurg. 2000 Nov;33(5):227-229. doi: 10.1159/000055959. PMID 11155057
- [Background] Sammartino M, Garra R, Sbaraglia F, De Riso M, Continolo N. Remifentanil in children. Paediatr Anaesth. 2010 Mar;20(3):246-55. doi: 10.1111/j.1460-9592.2009.03241.x. Epub 2010 Jan 21. PMID 20102527
- [Background] Kim SH, Stoicea N, Soghomonyan S, Bergese SD. Intraoperative use of remifentanil and opioid induced hyperalgesia/acute opioid tolerance: systematic review. Front Pharmacol. 2014 May 8;5:108. doi: 10.3389/fphar.2014.00108. eCollection 2014. PMID 24847273
- [Background] Abreu M, Aguado D, Benito J, Garcia-Fernandez J, Segura IA. Hyperalgesia and increased sevoflurane minimum alveolar concentration induced by opioids in the rat: a randomised experimental study. Eur J Anaesthesiol. 2015 Apr;32(4):232-41. doi: 10.1097/EJA.0000000000000188. PMID 25485881
- [Background] Weinbroum AA. Role of anaesthetics and opioids in perioperative hyperalgesia: one step towards familiarisation. Eur J Anaesthesiol. 2015 Apr;32(4):230-1. doi: 10.1097/EJA.0000000000000231. No abstract available. PMID 25747314
- [Background] Santonocito C, Noto A, Crimi C, Sanfilippo F. Remifentanil-induced postoperative hyperalgesia: current perspectives on mechanisms and therapeutic strategies. Local Reg Anesth. 2018 Apr 9;11:15-23. doi: 10.2147/LRA.S143618. eCollection 2018. PMID 29670398
- [Background] Guignard B, Bossard AE, Coste C, Sessler DI, Lebrault C, Alfonsi P, Fletcher D, Chauvin M. Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology. 2000 Aug;93(2):409-17. doi: 10.1097/00000542-200008000-00019. PMID 10910490
- [Background] Vinik HR, Kissin I. Rapid development of tolerance to analgesia during remifentanil infusion in humans. Anesth Analg. 1998 Jun;86(6):1307-11. doi: 10.1097/00000539-199806000-00033. PMID 9620525
- [Background] Lo C, Schwindt S, Sharma R, Dube R, Faraoni D, Steinberg BE, Brown S. Association Between Intraoperative Remifentanil Dosage and Postoperative Opioid Consumption in Adolescent Idiopathic Spine Surgery: A Retrospective Cohort Study. Anesth Analg. 2021 Oct 1;133(4):984-990. doi: 10.1213/ANE.0000000000005395. PMID 33555691
- [Background] Kaur M, Singh PM. Current role of dexmedetomidine in clinical anesthesia and intensive care. Anesth Essays Res. 2011 Jul-Dec;5(2):128-33. doi: 10.4103/0259-1162.94750. PMID 25885374
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Blaudszun G, Lysakowski C, Elia N, Tramer MR. Effect of perioperative systemic alpha2 agonists on postoperative morphine consumption and pain intensity: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2012 Jun;116(6):1312-22. doi: 10.1097/ALN.0b013e31825681cb. PMID 22546966
- [Background] Mason KP, Lerman J. Review article: Dexmedetomidine in children: current knowledge and future applications. Anesth Analg. 2011 Nov;113(5):1129-42. doi: 10.1213/ANE.0b013e31822b8629. Epub 2011 Aug 4. PMID 21821507
- [Background] Plambech MZ, Afshari A. Dexmedetomidine in the pediatric population: a review. Minerva Anestesiol. 2015 Mar;81(3):320-32. Epub 2014 May 14. PMID 24824958
- [Background] Wang Q, Chen C, Wang L. Efficacy and safety of dexmedetomidine in maintaining hemodynamic stability in pediatric cardiac surgery: a systematic review and meta-analysis. J Pediatr (Rio J). 2022 Jan-Feb;98(1):15-25. doi: 10.1016/j.jped.2021.05.008. Epub 2021 Jul 9. PMID 34252370
- [Background] Kiski D, Malec E, Schmidt C. Use of dexmedetomidine in pediatric cardiac anesthesia. Curr Opin Anaesthesiol. 2019 Jun;32(3):334-342. doi: 10.1097/ACO.0000000000000731. PMID 30893120
- [Background] Josephine C, Shariffuddin II, Chaw SH, Ng KWS, Ng KT. Hemodynamic Response of High- and Low-Dose Dexmedetomidine of Pediatric in General Anesthesia: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Asian J Anesthesiol. 2021 Mar 1;59(1):7-21. doi: 10.6859/aja.202103_59(1).0002. Epub 2021 Jan 21. PMID 33504143
- [Background] Gan L, Zhao X, Chen X. The Safety and Efficacy Evaluation of Dexmedetomidine for Procedural Sedation and Postoperative Behaviors in Pediatric Populations: A Systematic Review and Meta-analysis. Ann Pharmacother. 2022 Jan;56(1):16-26. doi: 10.1177/10600280211009845. Epub 2021 Apr 29. PMID 33913336
- [Background] Zhang SJ, Lai G, Griffis CA, Schiltz M, Aroke EN. alpha2-Adrenergic Receptor Agonist, an Attractive but Underused ERAS Component in Improving Fast-Track Recovery and Surgical Outcomes. AANA J. 2021 Dec;89(6):529-537. PMID 34809759
- [Background] Naduvanahalli Vivekanandaswamy A, Prasad Shetty A, Mugesh Kanna R, Shanmuganathan R. An analysis of the safety and efficacy of dexmedetomidine in posterior spinal fusion surgery for adolescent idiopathic scoliosis: a prospective randomized study. Eur Spine J. 2021 Mar;30(3):698-705. doi: 10.1007/s00586-020-06539-9. Epub 2020 Jul 21. PMID 32696258
- [Background] Schnabel A, Reichl SU, Poepping DM, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of intraoperative dexmedetomidine for acute postoperative pain in children: a meta-analysis of randomized controlled trials. Paediatr Anaesth. 2013 Feb;23(2):170-9. doi: 10.1111/pan.12030. Epub 2012 Oct 9. PMID 23043461
- [Background] Schnabel A, Meyer-Friessem CH, Reichl SU, Zahn PK, Pogatzki-Zahn EM. Is intraoperative dexmedetomidine a new option for postoperative pain treatment? A meta-analysis of randomized controlled trials. Pain. 2013 Jul;154(7):1140-9. doi: 10.1016/j.pain.2013.03.029. Epub 2013 Mar 27. PMID 23706726
- [Background] Tobias JD, Goble TJ, Bates G, Anderson JT, Hoernschemeyer DG. Effects of dexmedetomidine on intraoperative motor and somatosensory evoked potential monitoring during spinal surgery in adolescents. Paediatr Anaesth. 2008 Nov;18(11):1082-8. doi: 10.1111/j.1460-9592.2008.02733.x. PMID 18717802
- [Background] Anschel DJ, Aherne A, Soto RG, Carrion W, Hoegerl C, Nori P, Seidman PA. Successful intraoperative spinal cord monitoring during scoliosis surgery using a total intravenous anesthetic regimen including dexmedetomidine. J Clin Neurophysiol. 2008 Feb;25(1):56-61. doi: 10.1097/WNP.0b013e318163cca6. PMID 18303561
- [Background] Bagatini A, Volquind D, Rosso A, Trindade RD, Splettstosser JC. [Dexmedetomidine as adjuvant drug for wake-up test during scoliosis correction surgery: case report.]. Rev Bras Anestesiol. 2004 Apr;54(2):247-51. doi: 10.1590/s0034-70942004000200012. Portuguese. PMID 19471732
- [Background] Chen Z, Dai N, Lin S, Zhou G. Impact of Dexmedetomidine on Intraoperative Wake-Up Tests in Patients Undergoing Spinal Surgery. J Perianesth Nurs. 2018 Aug;33(4):448-452. doi: 10.1016/j.jopan.2016.07.009. Epub 2017 Apr 27. PMID 30077288
- [Background] Grape S, Kirkham KR, Frauenknecht J, Albrecht E. Intra-operative analgesia with remifentanil vs. dexmedetomidine: a systematic review and meta-analysis with trial sequential analysis. Anaesthesia. 2019 Jun;74(6):793-800. doi: 10.1111/anae.14657. Epub 2019 Apr 5. PMID 30950522
- [Background] Hwang W, Lee J, Park J, Joo J. Dexmedetomidine versus remifentanil in postoperative pain control after spinal surgery: a randomized controlled study. BMC Anesthesiol. 2015 Feb 24;15:21. doi: 10.1186/s12871-015-0004-1. eCollection 2015. PMID 25750586
- [Background] Wilson SH, Hellman KM, James D, Adler AC, Chandrakantan A. Mechanisms, diagnosis, prevention and management of perioperative opioid-induced hyperalgesia. Pain Manag. 2021 Apr;11(4):405-417. doi: 10.2217/pmt-2020-0105. Epub 2021 Mar 29. PMID 33779215
- [Background] Crawford MW, Hickey C, Zaarour C, Howard A, Naser B. Development of acute opioid tolerance during infusion of remifentanil for pediatric scoliosis surgery. Anesth Analg. 2006 Jun;102(6):1662-7. doi: 10.1213/01.ane.0000216036.95705.c2. PMID 16717305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited via investigator's review of medical records of their patients, approached by study team during inpatient or outpatient clinic visit, or referred to research team by their treating physician.
  Patients were enrolled from 12/20/2023 to 12/24/2024.
Period: Overall Study
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Full Range); unit: Years] — Mean Age in Years
  Years | 16 [14 to 19] | 17.2 [13 to 22] | 16.5 [13 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Count of Participants by Race/Ethnicity
  Participants
    Race/Ethicity: White | 6 | 6 | 12
    Race/Ethicity: Hispanic/Latino | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption (IV and PO in MME) on POD# 0 and 1
Description: Measure the median total opioid medications needed by the participants (IV and oral) after surgery on post operative days # 0 and 1.
Time Frame: Post Op Day# 0 and 1
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine
Number analyzed (Participants) | 7 | 6
MME
  MME POD 0 | 36.30 (71.90) [34.2 to 96.8] | 70.5 (66.98) [41.35 to 131.90]
  MME POD 1 | 57.5 [32.5 to 61.7] | 48 [41.9 to 54.1]

2. Secondary Outcome: Mean VAS Pain Score on POD# 0 and 1
Description: Measure the mean pain score of the participant on a visual analog pain scale. The VAS has two end points representing 0 ("no pain") and 10 ("worst pain ever"). It is reported at our institution as a number between 0 and 10.
Time Frame: Post Op Day# 0 and 1
Measure: Mean (Standard Deviation); unit: Visual Analog Pain Scale Score
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine
Number analyzed (Participants) | 7 | 6
Visual Analog Pain Scale Score
  VAS POD 0 | 3.39 (2.30) | 2.23 (1.40)
  VAS POD 1 | 3.32 (2.81) | 3.21 (0.98)

3. Secondary Outcome: Time From Skin Closure to Participant Being Able to Move Their Feet on Command (Mins)
Description: Measure the median time (mins) from completion of surgical skin closure to the participant being able to move their feet to command.
Time Frame: Intraoperative (day of surgery)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine
Number analyzed (Participants) | 7 | 6
Minutes | 14 [9 to 18] | 21.5 [10 to 30.75]

4. Secondary Outcome: Time From Skin Closure to Extubation
Description: Measure the median time (mins) from completion of surgical skin closure to extubation.
Time Frame: Intraoperative (day of surgery)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine
Number analyzed (Participants) | 7 | 6
Minutes | 15 [9.5 to 19] | 22 [11.75 to 31.75]

5. Primary Outcome: Total Opioid Consumption (IV and PO in MME) on POD# 0 and 1
Description: Measure the mean total opioid medications needed by the participants (IV and oral) after surgery on post operative days # 0 and 1.
Time Frame: Post Op Day# 0 and 1
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine
Number analyzed (Participants) | 7 | 6
MME
  MME POD 0 | 75.12 (71.58) | 88.93 (66.98)
  MME POD 1 | 54.38 (28.12) | 52.20 (27.40)

ADVERSE EVENTS:
Time Frame: From enrollment until inpatient discharge, up to 3 days.
Arm/Group | Propofol + Remifentanil | Propofol + Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
The study terminated early. Motor evoked potentials (MEP) is a monitor of spinal cord integrity, used to detect and prevent new neurological deficits in the context of spine surgery. Following anecdotally observed effects of some anesthetics interfering with MEP in patients undergoing scoliosis surgery, the surgeon involved in the study decided to pause enrollment and ultimately terminate the study early out of caution for patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT06096181/Prot_SAP_000.pdf